CLINICAL TRIAL: NCT01492855
Title: The Value of MRI in the Evaluation of Knees Suspected for Meniscal Lesions
Brief Title: Evaluation of MRI Diagnosed Meniscal Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ON-02-013-OSi
Record Dates: First submitted 2008-08-14; First posted 2011-12-15 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Meniscus Lesion
Keywords: Meniscal lesions; MRI; arthroscopic treatment
MeSH Terms: interventions — Arthroscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Operative treatment (Experimental)
  Interventions: Procedure: Arthroscopy
- Conservative treatment (Experimental)
  Interventions: Behavioral: Non-invasive treatment

INTERVENTIONS:
Procedure: Arthroscopy — Arthroscopy is offered for the patients who do not benefit from conservative treatment.
  Other Names: No other names.
  Arms: Operative treatment
Behavioral: Non-invasive treatment — All patients will receive information and supervised exercises by a physiotherapist.
  Other Names: No other names.
  Arms: Conservative treatment

SUMMARY:
The knee menisci are two semicircular fibrocartilaginous structures located between the articular cartilage surfaces of the femur and tibia in the medial and lateral joint compartments. The main functions of the menisci are shock absorption and load transmission in the knee, mainly through distribution of mechanical stress over a large area of the joint cartilage.

The hypothesis is that primarily older age, meniscal lesion and high pain score at baseline are associated with poorer outcome.

DETAILED DESCRIPTION:
Meniscal lesions are the most common source of disability of the knee with a reported incidence rate of up to 18 meniscal lesions per 10.000 subjects per year in Denmark. The meniscus may tear as a result of knee trauma or it may tear spontaneously due to aging and degenerative processes. Magnetic resonance imaging (MRI) is increasingly used in the diagnosis of meniscal lesions with documented high sensitivity and specificity. Meniscal lesion symptoms vary from reduction in knee function with decreased muscle strength and difficulties in performing strenuous activities involving knee flexion and rotation to pain, effusion locking and, giving way.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of meniscal lesion according to pain on weight-bearing activities, locking, normal stability, tenderness at medial and/or lateral joint line, normal X-ray
* Age > 18 years
* Able to understand Danish
* Able to sign an informed consent

Exclusion Criteria:

* Age < 18 years
* Unable to understand Danish
* Unable to sign an informed consent
* Unstable knee
* X-ray or MRI that shows other diagnoses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2008-01; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Investigation of improvement in KOOS subscale pain and symptoms | 12 months
  A multiple linear regression model is constructed to investigate which pre-treatment prognostic factors are associated to improvement in KOOS subscale pain and symptoms from baseline to follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Ole Simonsen, MD, Principal Investigator — Northern Orthopaedic Division
Locations (1):
- Northern Orthopaedic Division, Klinik Aalborg, Aalborg, Northern Jutland, Denmark